CLINICAL TRIAL: NCT06132334
Title: The Effects of Upper Extremity Aerobic Exercise Training on Exercise Capacity, Muscle Oxygen, and Physical Activity Level in Patients With Type 2 Diabetes
Brief Title: The Effects of Upper Extremity Aerobic Exercise Training in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Cardiopulmonary Physiotherapy and Rehabilitation, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gazi University63
Record Dates: First submitted 2023-10-22; First posted 2023-11-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type2diabetes
Keywords: Type 2 Diabetes Mellitus; Muscle oxygen; Oxygen consumption; Physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper extremity aerobic exercise training (Experimental): The training group will receive upper extremity aerobic exercise training on an arm ergometer accompanied by a physiotherapist for 6 weeks.
  Interventions: Other: Upper extremity aerobic exercise training
- Control Group (Sham Comparator): The control group will not be given any training for 6 weeks during the study period.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Upper extremity aerobic exercise training — Aerobic exercise training will be given to the training group on an arm ergometer 3 days in a week and 30-45 minutes a day for 6 weeks with the assistance of a physiotherapist. The training workload of aerobic exercise training will be applied at 50-80% of peak oxygen consumption or 60-80% of peak heart rate, dyspnea 3-4 points according to the Modified Borg Scale (MBS) or fatigue 4-6 points.
  Blood sugar measurement will be performed before exercise training. Individuals with a blood sugar result of >300 mg/dL will not be allowed to exercise that day.
  Arms: Upper extremity aerobic exercise training
Other: Control Group — The control group will not be given any training during the 6-week period. After the study, the treatment applied to the training group will also be applied to the control group in order to ensure that the patients in the control group are not ethically deprived of rehabilitation.
  Arms: Control Group

SUMMARY:
Type 2 diabetes (T2DM) is a metabolic disease characterized by chronic hyperglycemia that occurs as a result of any disorder in insulin secretion or insulin activity. Regular physical activity is important in preventing and managing this disease.

DETAILED DESCRIPTION:
T2DM causes significant mortality and morbidity, increases healthcare costs, and increases the risk of cardiovascular disease. Due to the rapid increase in the number of individuals with diabetes, preventing and controlling this disease and living with diabetes is important. In patients with T2DM, pulmonary functions decrease in relation to glycemic control and disease duration. Decrease in cardiorespiratory fitness can lead to cardiovascular mortality. Cardiovascular mortality increases as exercise capacity decreases. Although the determinants of exercise intolerance in diabetes are not fully understood, a number of abnormalities in pulmonary diffusion capacity, maximum cardiac output, blood oxygen capacity and skeletal muscle properties cause exercise tolerance. Peripheral factors such as skeletal muscles also affect exercise intolerance. Insufficient oxygen use in skeletal muscles is considered one of the causes of exercise intolerance in T2DM patients. To reduce the cardiovascular mortality rate and risk factors associated with cardiovascular disease, physical activity level is important in T2DM patients, as in all populations. Maintaining physical activity level plays a protective role against both T2DM and cardiovascular disease. But traditional exercise training guides generally focus on walking exercises. Because exercises in this form are frequently used in daily life activities. It is known that upper extremity movements are frequently used in daily living activities, and aerobic exercise using the upper extremities is thought to be safe and effective in these patients due to diabetic foot complications. There is no study in the literature investigating the effects of upper extremity aerobic exercise training in T2DM.

The primary aim of the study is to investigate the effects of upper extremity aerobic exercise training applied to T2DM patients on exercise capacity, muscle oxygenation and physical activity level.

The secondary aim of the study is to investigate its effects on upper extremity functional exercise capacity, dual task performance, respiratory functions, respiratory muscle strength and endurance, peripheral muscle strength, shortness of breath, fatigue, depression, anxiety, sleep and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2DM,
* Aged between 18-65 years,
* Able to walk and cooperate,
* Patients who volunteer to participate in the study.

Exclusion Criteria:

* Body mass index >40 kg/m2,
* A known lung disease,
* Serious neurological, neuromuscular, orthopedic, or other diseases affecting physical functions,
* Cognitive impairment that causes them to have difficulty understanding and following exercise test instructions,
* Having had any cardiac event or surgery in the last six months,
* Participated in a planned exercise program within the last three months,
* Uncontrolled hypertension,
* An acute pulmonary exacerbation within the last 4 weeks, have an acute upper or lower respiratory tract infection,
* Presence of diabetes complications such as nephropathy, retinopathy and severe neuropathy,
* Contraindications for exercise testing and/or exercise training according to the American College of Sports Medicine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption | through study completion, an average of 2 year
  Maximum exercise capacity will be assessed by symptom-limited cardiopulmonary exercise testing on a treadmill at gradually increasing speed and degree, and oxygen consumption will be measured during the test.
Muscle oxygenation | through study completion, an average of 2 year
  Before the cardiopulmonary exercise test and the 6-minute pegboard and ring test (6-PBRT), during and after the tests the muscle oxygenation will be measured by using a near-infrared spectroscopy device.
Physical activity level | through study completion, an average of 2 year
  A multi-sensor activity monitor will be used to assess the level of physical activity

SECONDARY OUTCOMES:
Upper extremity functional exercise capacity | through study completion, an average of 2 year
  It will be evaluated with a 6-minute pegboard and ring test. At the end of six minutes, the total number of rings inserted will be recorded in numbers.
Pulmonary function (Forced vital capacity (FVC)) | through study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | through study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | through study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | through study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | through study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, peak flow rate (PEF) will be evaluated.
Dual task performance | through study completion, an average of 2 year
  The test consists of 3 parts. Cognitive task, motor task and dual task will be evaluated. Patients will perform the Timed up and go (TUG) task as a single motor task. For the dual task, participants will be asked to perform the TUG test while counting down in increments of 3, starting from 100.As a single cognitive task, the individual will be asked to count down the specified number in increments of 3, while sitting comfortably in a quiet room, for the duration of the single task TUG. The total number of answers and the number of correct answers will be used to calculate the correct response rate as an indicator of cognitive performance during the dual task.
Respiratory Muscle Strength | through study completion, an average of 2 year
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria
Respiratory Muscle Endurance | through study completion, an average of 2 year
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load.
Peripheral muscle strength (N) | through study completion, an average of 2 year
  Shoulder flexion muscles and Quadriceps femoris muscle strength will be measured by using a hand-held dynamometer. This values is expressed in Newtons (N).
Dyspnea in daily life | through study completion, an average of 2 year
  "Modified Medical Research Council" dyspnea scale will be used to question dyspnea perception during activities. This scale is a 5-point scale based on rating various physical activities that increase shortness of breath. The lowest and highest values on this scale are as follows: Level 0 "No shortness of breath except strenuous exercise" and level 4 "Too breathless to leave the house or breathless while dressing or undressing."
Fatigue | through study completion, an average of 2 year
  Fatigue will be assessed with Fatigue Severity Scale (Turkish version). This scale includes 9 items and each item scores from 1 (strong disagreement) to 7 (strong agreement) point. Fatigue Severity Scale total score is calculates by deriving an arithmetic mean. Cut-score of over 4 means significant fatigue and higher score indicates more severe fatigue.
Anxiety and Depression | through study completion, an average of 2 year
  The Turkish version of the Hospital Anxiety and Depression Scale (HADS) will be used. HADS score ranges from 0-42. A high score indicates increased levels of anxiety and depression.
Sleep Quality | through study completion, an average of 2 year
  It will be evaluated with the Turkish version of the Epworth Sleepiness Scale (EDS). The scale is designed to evaluate the sleepiness level of individuals during the day and is widely used. Total score is between 0-24. The range specified for normal sleep tendency is considered to be 0-10 points. Sleep is disrupted with a score of 11 points or above.
Life quality | through study completion, an average of 2 year
  Quality of life will be evaluated with the Turkish adaptation of the Diabetes Quality of Life Scale (DQOL). The scale is calculated out of 0-100 points. High scores indicate good quality of life.
Diabetes symptoms | through study completion, an average of 2 year
  It will be evaluated with the Diabetes Symptoms Checklist Scale ((DSC-R).The total score and all subscale scores on the scale range from 0 to 5, with higher scores indicating greater symptom burden.
Dyspnea perception | through study completion, an average of 2 year
  Modified Borg Scale: The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath.
Peripheral muscle strength (%) | through study completion, an average of 2 year
  Shoulder flexion muscles and Quadriceps femoris muscle strength will be measured by using a hand-held dynamometer. This values is expressed as a percentage (%) of the expected value.
Upper extremity functional exercise capacity (percentage of the expected value (%)) | through study completion, an average of 2 year
  It will be evaluated with a 6-minute pegboard and ring test.The total number of rings each participant is expected to wear will be calculated. The percentage of the number of rings made relative to the expected value will be expressed as a percentage of the expected value (%).

CONTACTS AND LOCATIONS:
Overall Officials: Fidan YILMAZ, MSc, Study Chair — Gazi University; Ayşenur SARISAKALOĞLU, MSc, Principal Investigator — Gazi University; Serpil GÜLKAN, MD, Principal Investigator — Pursaklar State Hospital; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Clinic, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pan B, Ge L, Xun YQ, Chen YJ, Gao CY, Han X, Zuo LQ, Shan HQ, Yang KH, Ding GW, Tian JH. Exercise training modalities in patients with type 2 diabetes mellitus: a systematic review and network meta-analysis. Int J Behav Nutr Phys Act. 2018 Jul 25;15(1):72. doi: 10.1186/s12966-018-0703-3. PMID 30045740
- [Background] Kanaley JA, Colberg SR, Corcoran MH, Malin SK, Rodriguez NR, Crespo CJ, Kirwan JP, Zierath JR. Exercise/Physical Activity in Individuals with Type 2 Diabetes: A Consensus Statement from the American College of Sports Medicine. Med Sci Sports Exerc. 2022 Feb 1;54(2):353-368. doi: 10.1249/MSS.0000000000002800. PMID 35029593
- [Background] Amadid H, Johansen NB, Bjerregaard AL, Brage S, Faerch K, Lauritzen T, Witte DR, Sandbaek A, Jorgensen ME, Vistisen D. The role of physical activity in the development of first cardiovascular disease event: a tree-structured survival analysis of the Danish ADDITION-PRO cohort. Cardiovasc Diabetol. 2018 Sep 12;17(1):126. doi: 10.1186/s12933-018-0769-x. PMID 30208900
- [Background] Ibanez J, Izquierdo M, Arguelles I, Forga L, Larrion JL, Garcia-Unciti M, Idoate F, Gorostiaga EM. Twice-weekly progressive resistance training decreases abdominal fat and improves insulin sensitivity in older men with type 2 diabetes. Diabetes Care. 2005 Mar;28(3):662-7. doi: 10.2337/diacare.28.3.662. PMID 15735205
- [Background] Balducci S, Zanuso S, Nicolucci A, Fernando F, Cavallo S, Cardelli P, Fallucca S, Alessi E, Letizia C, Jimenez A, Fallucca F, Pugliese G. Anti-inflammatory effect of exercise training in subjects with type 2 diabetes and the metabolic syndrome is dependent on exercise modalities and independent of weight loss. Nutr Metab Cardiovasc Dis. 2010 Oct;20(8):608-17. doi: 10.1016/j.numecd.2009.04.015. Epub 2009 Aug 19. PMID 19695853
- [Background] Ur Rehman SS, Karimi H, Gillani SA, Ahmad S. Effects of supervised structured aerobic exercise training programme on level of Exertion, dyspnoea, VO2 max and Body Mass Index in patients with type 2 diabetes mellitus. J Pak Med Assoc. 2017 Nov;67(11):1670-1673. PMID 29171557
- [Background] Kirwan JP, Solomon TP, Wojta DM, Staten MA, Holloszy JO. Effects of 7 days of exercise training on insulin sensitivity and responsiveness in type 2 diabetes mellitus. Am J Physiol Endocrinol Metab. 2009 Jul;297(1):E151-6. doi: 10.1152/ajpendo.00210.2009. Epub 2009 Apr 21. PMID 19383872